CLINICAL TRIAL: NCT06918860
Title: Complications, Implant Survival and Functional Results After Surgical Treatment of Bone Metastases of Proximal Femur With Intramedullary Nail or Prosthetic Reconstruction
Brief Title: Analysis of Intramedullary Nail and Prosthetic Reconstruction After Surgical Treatment of Bone Metastases of Proximal Femur
Status: Recruiting | Type: Observational
Sponsor: Costantino Errani (Other)
Responsible Party: Sponsor-Investigator, Costantino Errani, Principal Investigator, Istituto Ortopedico Rizzoli
Organization: Istituto Ortopedico Rizzoli (Other)
Other Study IDs: BoneMetaProFe
Record Dates: First submitted 2025-03-26; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Bone Metastases
Keywords: bone metastases; proximal femur

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Male and female adult patients surgically treated between 01/01/2000 and 31/12/2023 in Rizzoli Orthopaedic Institute and in Massachusetts General Hospital.
  Interventions: Other: Analysis

INTERVENTIONS:
Other: Analysis — Analysis and review of imaging and clinical data

SUMMARY:
The investigators will collect data of patients treated surgically for impending or pathological fracture of the proximal femur due to bone metastases between 01/01/2000 and 31/12/2023 with IMN or THA or HHA or MegaTHA or Mega.

After pre-screening the databases of the respective sites, the investigators expect to find approximately a total of 600 patients. A review will be made from the medical records, radiological imaging, and histological data of partecipants.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adult patients surgically treated between 01/01/2000 and 31/12/2023 in Rizzoli Orthopaedic Institute and in Massachusetts General Hospital.
* Age ≥18 y (at the time of surgery)
* Patients with impending or pathological fracture due to bone metastases of the proximal femur (head/neck, intertrochanteric, subtrochanteric area).
* Patients who underwent either IMN or THA or HHA or Mega or MegaTHA.
* Patients with available clinical and imaging data.

Exclusion Criteria:

* Patients with pathological or impending fracture of proximal femur due to primary bone tumor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female adult patients surgically treated between 01/01/2000 and 31/12/2023 in Rizzoli Orthopaedic Institute and in Massachusetts General Hospital.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Analysis of implant survival | through study completion, an average of 1 year
  Assess the longevity associated with the different surgical treatments used for proximal femur bone metastases.
Analysis of complications | At baseline ( T0)
  Assess the post-operative complications associated with the different surgical treatments used for proximal femur bone metastases.
Analysis of functional score | 1 year
  Assess the functional score associated with the different surgical treatments used for proximal femur bone metastases.

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs Istituto Ortopedico Rizzoli, Bologna, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wedin R, Bauer HC. Surgical treatment of skeletal metastatic lesions of the proximal femur: endoprosthesis or reconstruction nail? J Bone Joint Surg Br. 2005 Dec;87(12):1653-7. doi: 10.1302/0301-620X.87B12.16629. PMID 16326880
- [Background] Errani C, Mavrogenis AF, Cevolani L, Spinelli S, Piccioli A, Maccauro G, Baldini N, Donati D. Treatment for long bone metastases based on a systematic literature review. Eur J Orthop Surg Traumatol. 2017 Feb;27(2):205-211. doi: 10.1007/s00590-016-1857-9. Epub 2016 Sep 20. PMID 27650452
- [Background] Araki N, Chuman H, Matsunobu T, Tanaka K, Katagiri H, Kunisada T, Hiruma T, Hiraga H, Morioka H, Hatano H, Asanuma K, Nishida Y, Hiraoka K, Okamoto T, Abe S, Watanuki M, Morii T, Sugiura H, Yoshida Y, Ohno T, Outani H, Yokoyama K, Shimose S, Fukuda H, Iwamoto Y. Factors associated with the decision of operative procedure for proximal femoral bone metastasis: Questionnaire survey to institutions participating the Bone and Soft Tissue Tumor Study Group of the Japan Clinical Oncology Group. J Orthop Sci. 2017 Sep;22(5):938-945. doi: 10.1016/j.jos.2017.05.012. Epub 2017 Jun 17. PMID 28629828